CLINICAL TRIAL: NCT04608396
Title: MERIT: A Randomized, Double-blind, Placebo-controlled Study of AXS-05 for Relapse Prevention in Treatment Resistant Depression
Brief Title: Mechanistic Evaluation of Response in TRD (MERIT)
Acronym: MERIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-05-TRD-201
Record Dates: First submitted 2020-10-07; First posted 2020-10-29 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: AXS-05; Treatment Resistant Depression; TRD; NMDA receptor; Refractory depression; Resistant depression; Depression; Major depression; Relapse prevention; Dextromethorphan; Bupropion
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AXS-05 (Experimental)
  Interventions: Drug: AXS-05
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 — AXS-05 taken daily for up to 52 weeks, until relapse.
  Arms: AXS-05
Drug: Placebo — Placebo taken daily for up to 52 weeks, until relapse.
  Arms: Placebo

SUMMARY:
To evaluate the relapse prevention of AXS-05 relative to placebo in subjects with treatment resistant depression (TRD).

This is a randomized, double-blind, placebo-controlled study to evaluate AXS-05 compared to placebo in delaying relapse of depressive symptoms in patients with TRD who are in stable remission after treatment with AXS-05.

ELIGIBILITY:
Key Eligibility Criteria:

* Ongoing symptoms of depression despite receiving treatment with two or more prior antidepressants during the current major depressive episode, prior to receiving AXS-05
* Agree to use adequate method of contraception for the duration of the study
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Relapse | Time from randomization to first relapse (up to 52 weeks)
  Assessed by clinician-rated scales.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, North Miami, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com